CLINICAL TRIAL: NCT05734001
Title: Rotational Thromboelastometry Versus Conventional Haemostatic Tests in Children With Decompensated Cirrhosis Undergoing Invasive Procedures:A Randomised Controlled Trial
Brief Title: Rotational Thromboelastometry Versus Conventional Haemostatic Tests in Children With Decompensated Cirrhosis Undergoing Invasive Procedures.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ILBS-DecompCirrhosis-01
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Haemostatic Tests (Active Comparator): Conventional Haemostatic Tests:
  1. If INR: > 2.5 FFP will be transfused at 15 ml/kg
  2. If Platelet Count is 20,000/mm3-50,000/mm3 RDPC will be transfused at 10 ml/kg
  3. If Fibrinogen < 80 mg/dl Cryoprecipitate will be transfused at 5 ml/kg
  Interventions: Diagnostic Test: Conventional Haemostatic Tests
- ROTEM Based tests (Experimental): The second group will undergo ROTEM based correction. ROTEM correction will be based on the following protocol :
  1. EXTEM CT > 80 sec - FFP will be transfused at 15 ml/kg MCF < 35 mm- Platelet will be transfused at 10 ml/kg
  2. FIBTEM MCF < 7 mm- Cryoprecipitate will be transfused at 5 ml/kg
  Interventions: Diagnostic Test: ROTEM Tests

INTERVENTIONS:
Diagnostic Test: ROTEM Tests — This group will undergo ROTEM based correction. ROTEM bcorrection will be based on the following protocol
  1. EXTEM CT > 80 sec - FFP will be transfused at 15 ml/kg MCF < 35 mm- Platelet will be transfused at 10 ml/kg
  2. FIBTEM MCF < 7 mm- Cryoprecipitate will be transfused at 5 ml/kg
  Arms: ROTEM Based tests
Diagnostic Test: Conventional Haemostatic Tests — To prevent bleeding during the procedure, one group will receive prophylactic transfusion of either FFP, Platelet or Cryoprecipitate based on the following protocol
  1. If INR: > 2.5 FFP will be transfused at 15 ml/kg
  2. If Platelet Count is 20,000/mm3-50,000/mm3 RDPC will be transfused at 10 ml/kg
  3. If Fibrinogen < 80 mg/dl Cryoprecipitate will be transfused at 5 ml/kg
  Arms: Conventional Haemostatic Tests

SUMMARY:
Decompesated Cirrhosis is charecterised by decreased synthesis of both procoagulants and anticoagulants along with thrombocytopenia and a delicate balance exists bleeding and thrombosis in this condition. There is increase in Prothrombin Time (PT) in this condition, consequently guidelines recommend correction of International Normalised Ratio (INR) and platelete count by transfusion of Fresh Frozen Plasma (FFP) and platelet transfusion before invasive procedures to prevent bleeding complications. However PT and platelet count are not ideal tests to guide transfusion strategies as they do not take into account the relative deficiency of anticoagulant factors. Furthermore, cirrhotic patients have an excess of von Willebrand factors and Factor VIII which are prothrombotic. So FFP and platelet transfusions based on PT and platelet count can actually lead to a prothrombotic state. Viscoelastic assays like ROTEM measure the haemostatic process in real time by detecting the resistance to movement of an oscillating pin by the clotting blood. It has three componenets-EXTEM, which measures the extrinsic coagulation pathway, INTEM, which measures the intrinsic pathway and FIBTEM which measures fibrinogen. Two parameters of EXTEM indicate FFP and platelet requirement and should be able to guide transfusion therapy. The first is Clottting Time (CT), that is the latency time between the formation of the test and the clot formation as the tracing reaches 2 mm of amplitude and the second is Maximum Clot Formation (MCF), that is the greatest vertical amplitude of the tracing. While CT helps in guiding FFP transfusion, MCF guides platelet transfusion. Fibrinogen requirement is guided by MCF values of FIBTEM.

The aim of this study will be to compare the transfusion requirement, efficacy and safety of ROTEM in guiding the use of FFP, Platelet and cryoprecipitate transfusion before invasive procedures in children with decompensated cirrhosis before invasive procedures.

Project title:Rotational Thromboelastometry versus conventional haemostatic tests in children with Decompensated Cirrhosis undergoing invasive procedures: A Randomised Controlled Trial

Student PI name: Dr Snigdha Verma

DETAILED DESCRIPTION:
a) Single centre Randomised Control Trial

(b) Methodology:

* Study population : Children aged6months-18 years with Decompensated Cirrhosis with histologic or image proven liver cirrhosis of any etiology with INR >2.5 and/or PLT count 20,000/mm3- 50,000/mm3 and who are listed for the following invasive procedure
* Low risk of bleeding

  1. Central venous cannulation
  2. Haemodialysis catheter
  3. Ascitic or Pleural tapping
  4. EVL
  5. EST

     High risk of bleeding
  6. TIPPS
  7. ERCP with sphicterotomy
  8. PCD Insertion
  9. Biopsies other than liver biopsy
* Study design:Randomised Control Trial
* Study period: 2 year: October 2022 to October 2024

STATISTICAL ANALYSIS: Sample size calculation for the RCT

* Appropriate statistical test for correlation analysis will be applied
* Assuming a 20% difference in the average transfusion requirements of the two groups based on a previous study, assuming a 5% alpha error and power of 90% along with an expected dropout rate of 10%, we got a sample size of 90 (45 patients in each arm) and 1/3rd patients of this would be for Liver Biopsy.

Intervention :

* Children with decompensated cirrhosis listed for invasive procedures and with deranged INR between >2.5and/or deranged platelet count between 20,000/mm3-50,000/mm3 will be included in the study and will undergo block randomization into two groups. To prevent bleeding during the procedure, one group will receive prophylactic transfusion of either FFP, Platelet or Cryoprecipitate based on the following protocol

  1. If INR: > 2.5 FFP will be transfused at 15 ml/kg
  2. If Platelet Count is 20,000/mm3-50,000/mm3 RDPC will be transfused at 10 ml/kg
  3. If Fibrinogen < 80 mg/dl Cryoprecipitate will be transfused at 5 ml/kg The second group will undergo ROTEM based correction. ROTEM bcorrection will be based on the following protocol

  <!-- -->

  1. EXTEM CT > 80 sec - FFP will be transfused at 15 ml/kg MCF < 35 mm- Platelet will be transfused at 10 ml/kg
  2. FIBTEM MCF < 7 mm- Cryoprecipitate will be transfused at 5 ml/kg

Following correction, the procedure will be done in both the groups. Patients randomised in the ROTEM group will undergo repeat ROTEM and INR, Platelet, Fibrinogen testing (depending on the component transfused), post the procedure, to look at the correction achieved. Similarly, patients randomised in the conventional group will undergo repeat INR, Platelet,fibrinogen testing depending on the component transfused.

Patients will be followed for 24 hours indoors for any evidence of bleeding or transfusion reaction. Significant Bleeding have been defined as fall in Hb by 3 g/dl in 24 hours and /or hypotension CBC will be repeated at 24 hours, to look for any fall. Transfusion reactions that will be looked for Early (within 24 hours of transfusion) Severe allergic reaction - Acute hypotension, lower airway obstruction with urticaria, angioedema or generalized pruritis Transfusion related acute lung injury-New acute lung injury within 6 hours of a transfusion; Hypoxemi with PaO2/FiO2 < 300 mm Hg ( or O2 < 90%) and bilateral Chest X ray infilterates with lack of other risk factors for pulmonary edema.

Transfusion associated circulatory overload- Acute onset of congestive heart failure as a direct result of blood transfusion with

1. Dyspnea, orthopnea, bilateral rales with hypoxia or
2. Systolic Hypertension, tachycardia, jujgular venous distension, pedal edema with A) X rays with bilateral basilar infiltrates or B) Hypoxemia (< 90% saturation on room air)

Patient will be followed up in OPD after 5 days to look for any late transfusion reaction Delayed reactions looked forwill be Delayed hemolytic transfusion reaction Hemolysis after 24 hours with anemia, DCT positivity, spherocytes on peripheral smear Monitoring and assessment:The amount of total blood components (FFP, Platelet, Cryoprecipitate) transfused in each group will be assessed, along with the amount of individual components transfused. The bleeding episodes will be assessed by fall in Hb or blood pressure in each group, as will be the transfusion reactions (Acute respiratory distress syndrome, Transfusion related acute lung injury, Heart failure or majortransfusion reactions.

STATISTICAL ANALYSIS: Sample size calculation for the RCT Appropriate statistical test for correlation analysis will be applied

- Adverse effects: Patientsreceiving transfused blood componets based on ROTEM or conventional methods will be monitored for clinically significant bleeding till 24 hours post procedure. Transfusion reactions in the form of ARDS, TRALI will be looked for.

- Stopping rule: Interim analysis will be done after 20 patients. If significant increase in the bleeding rate or transfusion reactions in the ROTEM group, trial will be stopped

e) Ethical issues in the study and plans to address these issues: The transfusion requirement in the ROTEM group is expected to reduce as compared to the transfusion requirement in the Conventional group. This is expected to reduce the number of transfusion reactions and the cost of therapy in the ROTEM group. The additional of cost of doing ROTEM tests is expected to be mitigated by the reduction in cost from decreased transfusion requirement and decreased transfusion reaction.

ELIGIBILITY:
Inclusion Criteria:

* Children 6m- 18years of age
* Histologic or image proven liver cirrhosis of any etiology
* Listed for an invasive procedure Procedures 1. Central venous cannulation 2. Haemodialysis catheter 3. Ascitic or Pleural tapping 4. EVL/EST 5. TIPPS 6. ERCP with sphicterotomy 7. PCD Insertion 8. Biopsies other than liver biopsy : INR >2.5 and/or PLT count 20,000/mm3- 50,000/mm3 9. Those listed for Liver Biopsy: INR >2 and/or PLT count 20-50,000/mm3

Exclusion Criteria:

* Anti platelet or anti coagulant therapy in the previous 7 days
* Patients with clinical evidence of DIC and/or active bleeding
* Hemodialysis in the past 7 days

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The amount of total component transfused (ml/kg) will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis | 1 day

SECONDARY OUTCOMES:
The amount of FFP (ml/kg) transfused will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis | 1 day
The amount of Platelet (ml/kg) transfused will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis. | 1 day
The amount of cryoprecipitate (ml/kg) transfused will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis | 1 day
The bleeding rate will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis | 5 days
The rate of transfusion reactions will be significantly less in Rotational Thromboelastometry guided therapy versus Conventional therapy for invasive procedures in children with cirrhosis | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India